CLINICAL TRIAL: NCT06071312
Title: Fecal Microbiota Transplantation in Patients With Recurrent Clostridioides Cifficile Infection and Ulcerative Colitis: Single Infusion Versus Sequential Approach
Brief Title: FMT in Patients With Recurrent CDI and Ulcerative Colitis: Single Infusion Versus Sequential Approach
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, IANIRO GIANLUCA, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5183
Record Dates: First submitted 2023-10-03; First posted 2023-10-06 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Clostridium Difficile; Ulcerative Colitis
Keywords: Ulcerative Colitis; Clostridium difficile; Fecal microbiota transplantation
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, open-label, single-center trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- . Single FMT (Experimental): Patients enrolled in this arm will receive a single infusion of donor FMT
  Interventions: Biological: single FMT
- Sequential FMT (Active Comparator): Patients enrolled in this arm will receive sequential infusions of donor FMT
  Interventions: Biological: sequential FMT

INTERVENTIONS:
Biological: single FMT — This intervention is represented by the administration, in the recipients' gut, of healthy donor microbiota through a single infusion of FMT
  Arms: . Single FMT
Biological: sequential FMT — This intervention is represented by the administration, in the recipients' gut, of healthy donor microbiota through multiple infusions of FMT (sequential approach)
  Arms: Sequential FMT

SUMMARY:
Clostridioides difficile infection (CDI) is the most frequent cause of infectious diarrhea in hospitalized patients and is responsible for 20-30 % of antibiotic-associated diarrhea cases. Inflammatory bowel diseases (IBD) are associated with an higher prevalence, recurrence and severity of CDI. The prevalence of recurrent CDI in patients with IBD is 2.5 to 8 times higher than in the general population, with a cumulative lifetime risk of 10 %. The higher risk to the development of CDI in patient with IBD is directly related to the microbiome alterations that are associated with this chronic disoder. Moreover, the use of antibiotics to cure CDI further worsens the gut microbiota, triggering potentially a self-maintaining cycle and predisposes such patients to a higher risk of recurrence. In these patients, CD superinfection is associated, with an increased rate of hospitalization, length of stay, the need to modify the treatment to the underlying disease, the increase rate of colectomy, there higher mortality rate, with a net increase of health costs.

Nowadays, as emerged by several studies FMT has been established as a valid treatment option against recurrent CDI (rCDI), and it is recommended by international guidelines.

Unfortunately, most FMT studies for rCDI have excluded patients with IBD. Recent evidence suggests that FMT is effective in patients with ulcerative colitis (UC) and concomitant rCDI, both in the treatment of the infection and in the improve of disease activity. To date, most studies evaluated the efficacy of single infusion of FMT in these patients.

Preliminary data from our group suggest that a sequential approach (i.e., repeated fecal infusions) may increase the efficacy of FMT in this population. Indeed, in 18 patients with IBD, single infusion fecal resulted in eradication of rCDI in 60% of cases, whereas this outcome was achieved in 89% of cases using a sequential approach. Similar data have been demonstrated in a retrospective study by Fischer and colleagues. However, more studies are advocated to confirm these results.

Therefore, our study aim to compare the efficacy of single FMT vs. sequential in the eradication of rCDI in patients with UC.

DETAILED DESCRIPTION:
Clostridioides difficile infection (CDI) is the most frequent cause of infectious diarrhea in hospitalized patients and is responsible for 20-30 % of antibiotic-associated diarrhea cases. Inflammatory bowel diseases (IBD) are associated with an higher prevalence, recurrence and severity of CDI. The prevalence of recurrent CDI in patients with IBD is 2.5 to 8 times higher than in the general population, with a cumulative lifetime risk of 10 %. The higher risk to the development of CDI in patient with IBD is directly related to the microbiome alterations that are associated with this chronic disoder. Moreover, the use of antibiotics to cure CDI further worsens the gut microbiota, triggering potentially a self-maintaining cycle and predisposes such patients to a higher risk of recurrence. In these patients, CD superinfection is associated, with an increased rate of hospitalization, length of stay, the need to modify the treatment to the underlying disease, the increase rate of colectomy, there higher mortality rate, with a net increase of health costs.

Nowadays, as emerged by several studies FMT has been established as a valid treatment option against recurrent CDI (rCDI), and it is recommended by international guidelines.

Unfortunately, most FMT studies for rCDI have excluded patients with IBD. Recent evidence suggests that FMT is effective in patients with ulcerative colitis (UC) and concomitant rCDI, both in the treatment of the infection and in the improve of disease activity. To date, most studies evaluated the efficacy of single infusion of FMT in these patients.

Preliminary data from our group suggest that a sequential approach (i.e., repeated fecal infusions) may increase the efficacy of FMT in this population. Indeed, in 18 patients with IBD, single infusion fecal resulted in eradication of rCDI in 60% of cases, whereas this outcome was achieved in 89% of cases using a sequential approach. Similar data have been demonstrated in a retrospective study by Fischer and colleagues. However, more studies are advocated to confirm these results.

Therefore, our study aim to compare the efficacy of single FMT vs. sequential in the eradication of rCDI in patients with UC.

The extended aims of our study are:

* To compare the efficacy of single FMT versus sequential FMT in eradicating rCDI in patients with UC at 8 weeks after the end of treatment.
* To compare the efficacy of single FMT versus sequential FMT in the eradication of rCDI in patients with UC in the short term (1-4 weeks after the end of treatment).
* To evaluate the safety of the two treatments.
* To evaluate any changes in the microbiota following treatment.
* To assess disease activity of UC by clinical scores (partial Mayo score) at 8 weeks.

The investigators will carry out a randomized, controlled, open-label, single-clinical trial of single FMT vs sequential FMT in patients with active UC with concomitant rCDI, will be recruited among those referred to the gastroenterology unit of the Fondazione Policlinico Universitario "A. Gemelli". Patients with all inclusion criteria and none of the exclusion criteria (detailed in the specific section of this website) will be considered for this study.

Before randomization, demographic data will be collected by the gastroenterology staff.

Moreover, patients will be requested to give stool samples to be collected in a sterile, sealed container and stored at -80°C for metagenomic assessment of gut microbiome by the microbiology staff.

After baseline assessments, patients will be randomly assigned to one of the following treatment arms:

* Single FMT (Si-FMT);
* Sequential FMT (Se-FMT), consisting of 3 fecal infusions, each 3-6 days apart, within 18 days after randomization.

Each patient will undergo FMT procedure through colonoscopy under sedation; Fecal infusates will be delivered through the operative of the colonoscope, using 50-mL syringes.

Patients in the Si-FMT and Se-FMT arms will receive frozen feces from a healthy non related donor following the protocols suggested by the international guidelines. Patients in the Se-FMT arm will receive frozen feces from the same donor.

The selection of stool donors will be performed by the gastroenterology staff following protocols previously recommended by international guidelines and according the new recommendation imposed by the reorganization of fecal microbiota transplant during the COVID-19 pandemic.

The assignment of fecal infusates from healthy donors to patients will be done randomly, without any specific recipient- donor match, as this is not recommended by international guidelines All fecal infusates will be manufactured in the microbiology unit of our hospital. Only frozen feces will be used. Preparation of frozen feces will follow protocols from international guidelines.

Follow-up visits will be performed by physicians from the gastroenterology unit. All patients will be followed up for 2 months after the end of treatments. Follow- up visits will be scheduled at week 1, week 4, and week 8, after the end of treatments.

At each visit the following assessments will be performed: 1) collection of a stool sample for C. difficile toxin evaluation; 2) collection of a stool sample for metagenomic analysis of the gut microbiota; 3) clinical evaluation of disease activity; and 4) recording of adverse events.

Study Outcomes are detailed in the specific section of this website.

The statistical analysis will be performed both on an intention-to-treat and per- protocol basis. Differences among groups will be assessed with a two tailed Wilcoxon-rank sum test for continuous data and with Fisher's exact probability test (using two-tailed P-values) for categorical data. Differences in cure percentages will be determined with Fisher's exact test (with two-tailed P values). Microbiome analysis will be performed with shotgun sequencing techniques. For microbiome analysis statistical differences between group means will be calculated using a two-tailed Wilcoxon-Rank Sum Test, through the R statistical software package (R Core Team, Vienna, Austria).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Active UC (partial Mayo score ≥2);
* Relapsing infection of C. difficile;
* Ability to express consent for inclusion in the study.
* Indication, in the clinical practice setting, for fecal microbiota transplantation from a healthy donor for recurrent CDI

Exclusion Criteria:

* Age < 18 years;
* Other gastrointestinal infections, excluding C. difficile;
* Known gastrointestinal diseases, other than UC, in active stage (e.g., infectious gastroenteritis, celiac disease, irritable bowel syndrome, chronic pancreatitis, bile acid diarrhea, etc.);
* Previous colon surgery or skin ostomy packing;
* Food allergies;
* Current or recent (<2 weeks) therapy with drugs that may alter the microbiota (e.g., systemic antimicrobials, probiotics, proton pump inhibitors, immunosuppressants, metformin), except antibiotics against C. difficile;
* Heart failure or heart disease with FE ≤ 30 %;
* Severe respiratory failure;
* Psychiatric disorders;
* Pregnancy and lactation;
* Inability to provide informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-09-23 (Actual); Primary Completion 2025-09-24 (Estimated); Study Completion 2025-09-24 (Estimated)

PRIMARY OUTCOMES:
Number of UC patients who will obtain the eradication of rCDI 8 weeks after treatments (single FMT vs sequential FMT) | 2 months
  The investigators will compare the number of participants who will obtain the eradication of rCDI (assessed by C. difficile toxin exam) 8 weeks after treatments (single FMT vs sequential FMT)

SECONDARY OUTCOMES:
Number of UC patients who will obtain the eradication of rCDI 1 - 4 weeks after treatments (single FMT vs sequential FMT) | 1 months
  The investigators will compare the number of participants who will obtain the eradication of rCDI (assessed by C. difficile toxin exam) 1 - 4 weeks after treatments (single FMT vs sequential FMT).
Evaluation of changes in recipients' microbiome after treatments, at each time point. | 2 months
  The investigators will evaluate the characteristics of recipients' microbiome, assessed by metagenomics analysis, 1,4 and 8 weeks days after treatments, compared to baseline and donors' microbiome.
Evaluation of Ulcerative Colitis activity | 2 months
  The investigators will evaluate the clinical characteristics of ulcerative colitis, assessed by partial Mayo score, 1,4 and 8 weeks after treatments.
Evaluation of the safety of the two treatments | 2 months
  The investigators will record any adverse events (mild to severe) reported by participants, after treatments at each timepont.

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Ianiro, MD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Digestive Disease Center, Fondazione Policlinico Univesitario A. Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available to other researchers
Supporting Information: Study Protocol
Time Frame: data will be available after the completion of the study, for 5 years
Access Criteria: Data will be given upon request to the PI